CLINICAL TRIAL: NCT02821143
Title: The Impact of Telemedicine to Support Palliative Care Resident in Nursing Home: a Cluster Randomized Control Study.
Brief Title: The Impact of Telemedicine to Support Palliative Care Resident in Nursing Home
Acronym: TELESM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Realization not possible
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/15/7835
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Palliative Care
Keywords: Telemedicine; Nursing Home; Hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Every patient identified as belonging to a palliative care after the inclusion criteria will receive intervention with a follow-up with Telemedicine consultation
  Interventions: Other: Telemedicine consultation
- Control group (Other): Every patient identified as belonging to a palliative care after the inclusion criteria will receive Usual palliative care
  Interventions: Other: usual palliative care

INTERVENTIONS:
Other: usual palliative care — Residents in the control group will receive usual palliative care usually delivered in their nursing homes , according to the habits of the healthcare team and their physician.
  Arms: Control group
Other: Telemedicine consultation — Establishment of an initial multiprofessional Telemedicine consultation involving a palliative care physician and / or geriatrician, and other physician coordinator of nursing homes, health care team and if possible the patient's treating physician (patient and / or family may participate if they want to).
  The aim is to define and formalize:
  * Aid to collection and application of advanced directives according to Leonetti Act if the resident is able to do so, or collection of confidence personal choices.
  * Definition of the objectives of care and patient's life and therapeutic adaptation with a focus on pain and uncomfortable symptoms.
  * Access to a mobile team of palliative care or geriatric hospitalization at home, a hospice network, if the patient's situation requires.
  * In case of medical worsening :
  Possibility of access to consultations and use of emergency by tele-expertise or decision support within a maximum period of 72 hours, with the same objectives that above.
  Arms: Intervention group

SUMMARY:
Investigators hypothesize that telemedicine may be an effective tool to improve palliative care in nursing home, by providing on-site specialized and interprofessional consultation. The objective of this study is to assess the impact of telemedicine in decreasing the rate of hospitalization, compared with usual care, in nursing home resident with palliative care needs.

DETAILED DESCRIPTION:
According to current statistics, approximately 12 % of all deaths in France occur in Nursing Home, with the number over 25% in USA. With the ageing of the population, this rate is expected to dramatically increase in the next years, to reach 40% in USA in 2020. Yet, there is some evidence that palliative care is often inadequate in Nursing Home: there is a difficulty to recognize residents who might benefit palliative care and their needs, an underassessment and under-treatment of pain and other end-of-life symptoms, and frequent burdensome treatments and hospitalizations. Several programs including palliative care consult service (with outside consultant), Nursing Home-based palliative care or Nursing Home-hospice partnerships, have succeeded in delivering high-quality palliative care in Nursing Home. But, to our knowledge, no studies examined the benefit of telemedicine for palliative care in nursing home.

During a 6 month-inclusion period, residents with palliative care needs will be included in both arms. In the intervention group, Telemedicine consultations involving Nursing Home staff and the palliative and/or geriatric unit from the University Hospital, will be organized systematically at inclusion and during the follow-up if needed. In both groups, hospitalizations and emergency hospitalizations, quality of life of the resident, satisfaction of the nursing home staff and health costs will be recorded during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Residents with palliative care needs:

  * Diagnosis of advanced or terminal disease: advanced cancer, advanced congestive Hearth Failure, end-stage pulmonary disease, end-stage hepatic disease, end-stage neurologic disease, other end-stage medical diagnosis.
  * ≥ A unplanned acute hospital episodes within the past 6 months
  * Activity of daily life ≤ 1 and/or bed/chair ridden residents for at least 30 days.
  * Weight loss ≥ 10% of body weight in the last 6 months.
  * The " surprise question " approach: " Would I be surprised if this patient died within the next 6-12 months? "
* Informed and written consent by the patient or the legal representative or the reliable person when appropriate.
* General Practitioner agreement.

Exclusion Criteria:

* No agreement of study participation of patients or legal representative or the reliable person when appropriate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tele-expertise effectiveness on hospitalization rates | through the end of study (24 months)
  Evaluation by proportion of subject hospitalized at least one time during follow-up period

SECONDARY OUTCOMES:
Evaluation of tele-expertise effectiveness on emergency | through the end of study (24 months)
  Emergency hospitalization rates with proportion of subject hospitalized in emergency at least one time during follow-up period
Evaluation of tele-expertise effectiveness on last 15 days of life hospitalization rates | through the end of study (24 months)
  proportion of subject hospitalized in the last 15 days of life at least one time during follow-up period
Patient quality of life | 1 month after inclusion
  Assessed by Palliative Care Outcome Scale (PCOS)
Patient quality of life | 3 month after inclusion
  Assessed by Palliative Care Outcome Scale (PCOS)
Patient quality of life | 6 month after inclusion
  Assessed by Palliative Care Outcome Scale (PCOS)
Patient quality of life | Last patient's 3 days of life
  Assessed by Palliative Care Outcome Scale (PCOS)
Caregivers satisfaction | through the end of study (24 months)
  Assessed through a satisfaction survey
Economical evaluation | through the end of study (24 months)
  Evaluation of taking care costs with french social security scheme data

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Sourdet, MD, Principal Investigator — University Hospital of Toulouse

IPD SHARING:
Plan to Share IPD: No